CLINICAL TRIAL: NCT02929277
Title: Protection Against Allergy: Study in Rural Environment - Part IV
Acronym: PATURE IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R/2012/47
Record Dates: First submitted 2016-09-30; First posted 2016-10-11 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2016-10

CONDITIONS: Asthma; Atopy
Keywords: farm children; non-farm children
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Other)
  Interventions: Other: blood sampling, skin prick tests, assesment of atopic dermatitis, questionnaires

INTERVENTIONS:
Other: blood sampling, skin prick tests, assesment of atopic dermatitis, questionnaires

SUMMARY:
PASTURE is a birth cohort of children born to farm and non-farm women from rural areas across Europe. Five study centres Austria, Germany, Switzerland, France and Finland enrolled 1133 children (farmers in about half of the children) to study the origins of asthma and atopy and to develop potential preventive strategies.

Previous results show a protective effect of farm exposure on allergic risk by livestock contacts and microbial exposures and by raw cow milk consumption in early age.

PASTURE Part IV is the 10-year follow up of this birth cohort. The primary objective is to characterize the allergic phenotype between 6 and 10 years old (asthma and allergic rhinitis) and to explain how early age exposures and particularly milk products consumption contribute in the process of allergic illness in childhood. A focus on the characterization of the protective biologically active components in raw milk and identification of immunological mechanisms are involved.

ELIGIBILITY:
Inclusion Criteria:

* PATURE IV is a birth cohort. All children enrolled at the beginning and who still agree to participate will be included at 10-year follow-up.

Exclusion Criteria:

-

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05-06 (Actual)

PRIMARY OUTCOMES:
Asthma | 10 years old
Rhinitis | 10 years old
Atopic Dermatitis | 10 years old
Food Allergy | 10 years old
Skin prick tests | 10 years old
Specific Immunoglobulin E (IgEs) | 10 years old
Blood cytokine profiles | 10 years old

REFERENCES:
- [Result] Chauveau A, Dalphin ML, Mauny F, Kaulek V, Schmausser-Hechfellner E, Renz H, Riedler J, Pekkanen J, Karvonen AM, Lauener R, Roduit C, Vuitton DA, von Mutius E, Dalphin JC; PASTURE Study Group. Skin prick tests and specific IgE in 10-year-old children: Agreement and association with allergic diseases. Allergy. 2017 Sep;72(9):1365-1373. doi: 10.1111/all.13148. Epub 2017 Apr 12. PMID 28235151
- [Result] Chauveau A, Dalphin ML, Kaulek V, Roduit C, Pugin A, von Mutius E, Vuitton DA, Dalphin JC. Disagreement between Skin Prick Tests and Specific IgE in Early Childhood. Int Arch Allergy Immunol. 2016;170(2):69-74. doi: 10.1159/000446776. Epub 2016 Jul 26. PMID 27454436